CLINICAL TRIAL: NCT01769664
Title: A Randomized, Double-Blind, Multiple-Site, Placebo-Controlled, Parallel Design Study Comparing Clindamycin 1%/Benzoyl Peroxide 5% Topical Gel (Taro Pharmaceuticals Inc.) to Duac® Topical Gel Clindamycin 1%/Benzoyl Peroxide 5% (Stiefel) in the Treatment of Acne Vulgaris
Brief Title: A Study Comparing Clindamycin 1%/Benzoyl Peroxide 5% Topical Gel to Duac® Topical Gel in the Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLBG 1209
Record Dates: First submitted 2012-10-11; First posted 2013-01-17 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Acne Vulgaris
Keywords: Acne vulgaris; Clindamycin 1%/Benzoyl Peroxide 5% Topical Gel; Duac® Topical Gel
MeSH Terms: conditions — Acne Vulgaris | interventions — Clindamycin; Benzoyl Peroxide; Gels

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Clindamycin 1%/Benzoyl Peroxide 5% Topical Gel (Experimental): Clindamycin 1%/Benzoyl Peroxide 5% Topical Gel (Taro Pharmaceuticals Inc.)
  Interventions: Drug: Clindamycin 1%/Benzoyl Peroxide 5% Topical Gel
- Duac® Topical Gel (Active Comparator): Duac® (Clindamycin 1%/Benzoyl Peroxide 5%) Topical Gel (Stiefel)
  Interventions: Drug: Duac® Topical Gel
- Placebo Topical Gel (Placebo Comparator): Placebo (Vehicle) Topical Gel (Taro Pharmaceuticals Inc.)
  Interventions: Drug: Placebo Topical Gel

INTERVENTIONS:
Drug: Clindamycin 1%/Benzoyl Peroxide 5% Topical Gel — Clindamycin 1%/Benzoyl Peroxide 5% Topical Gel (Taro Pharmaceuticals Inc.) applied once a day in the evening for 77 days (11 weeks)
  Arms: Clindamycin 1%/Benzoyl Peroxide 5% Topical Gel
Drug: Duac® Topical Gel — Duac® (Clindamycin 1%/Benzoyl Peroxide 5%) Topical Gel (Stiefel) applied once a day in the evening for 77 days (11 weeks)
  Arms: Duac® Topical Gel
Drug: Placebo Topical Gel — Placebo (Vehicle) Topical Gel (Taro Pharmaceuticals Inc.) applied once a day in the evening for 77 days (11 weeks)
  Arms: Placebo Topical Gel

SUMMARY:
The objective of this study is to compare the relative efficacy and safety of the test formulation Clindamycin 1%/Benzoyl Peroxide 5% Topical Gel (Taro Pharmaceuticals Inc.) to the marketed formulation Duac® Topical Gel (Clindamycin 1%/Benzoyl Peroxide 5%) (Stiefel) in the treatment of the inflamed lesions of acne vulgaris. Both the test and reference formulations will also be compared to a placebo formulation to test for superiority.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating female, between 12 and 40 years of age with a clinical diagnosis of acne vulgaris.
* Signed informed consent form. For a minor, the parent or legal guardian will sign the consent form and patient will sign assent to participate form.
* If female of child-bearing potential, prepare to abstain from sexual intercourse or use a reliable method of contraception during the study. Patients on hormonal contraceptives must have been on the same for three months prior to baseline visit and continue throughout the duration of the study.
* Have facial acne with 20 or more facial inflammatory lesions and 25 or more non-inflammatory lesions and 2 or less nodulocystic lesions and have an Investigator Global Assessment score of 2, 3 or 4.
* Willing to comply with the study requirements and restrictions including refraining from the use of all other topical acne medications or antibiotics during the treatment period.

Exclusion Criteria:

* Patient has more than 2 facial nodular lesions.
* Patient has active cystic acne.
* Patient has acne conglobata.
* Patients with excessive facial hair that would interfere with the diagnosis or assessment of acne.
* Patients with tatoos or excessive facial scarring that may interfere with the evaluation of the patient's acne.
* Patients with active facial sunburn, peeling due to sunburn and patients who will be exposed to excessive sunlight during the study.
* Any skin condition other than acne vulgaris that would interfere with the evaluation of the patient's acne.
* Females who are pregnant, lactating or likely to become pregnant during the study.
* Patients with a history of or active colitis other than irritable bowel syndrome.
* History of allergy or hypersensitivity to Clindamycin, Lincomycin or benzoyl peroxide or history of any drug hypersensitivity or intolerance which would compromise the patient's safety or the study.
* Significant history or current evidence of chronic infectious disease, system disorder, organ disorder or other medical condition that would place the patient at undue risk by participation.
* Use on the face within 1 month prior to screening/baseline or during the study of the following: cryodestruction or chemodestruction, dermabrasion, photodynamic therapy, acne surgery, intralesional steroids, x-ray therapy.
* Use of the following within 1 month prior to screening/baseline: spironolactone, systemic steroids, systemic antibiotics, systemic treatment for acne vulgaris (other than oral retinoids which require a 6 month washout), systemic anti-inflammatory agents.
* Use of oral isotretinoin (Accutane®) or oral retinoids within 6 months, or therapeutic vitamin A supplements greater than 10,000 units/day.
* Use within 2 weeks prior to screening/baseline of the following: topical steroids, topical retinoids, topical acne treatments including over-the-counter preparations, topical anti-inflammatory agents, medicated cleansers, topical antibiotics.
* Receipt of any drug as part of a research study within 30 days.
* Female patients taking hormonal contraceptives or oral estrogen for less than 3 months and those that plan to change the dosage regimen during the course of the study.
* Previous participation in this study.
* Employees of the investigator or research center or their immediate family members.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 650 (Actual)
Dates: Start 2012-09; Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Bioequivalence of test gel to reference gel | Week 11 (study day 77)
  Bioequivalence will be determined by evaluating the mean percent change from baseline to week 11 in the number of inflammatory lesions.

SECONDARY OUTCOMES:
Superiority against placebo | Week 11 (study day 77)
  The superiority of the test and reference against the placebo will be tested for the mean percent reduction in inflamed lesion count at week 11.